CLINICAL TRIAL: NCT06533423
Title: Effect of a Self-Management Intervention for Patients Newly Diagnosed With Inflammatory Arthritis: Study Protocol for a Randomized Controlled NISMA Trial
Brief Title: Effect of a Self-Management Intervention for Patients Newly Diagnosed With Inflammatory Arthritis: The NISMA Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Bente Appel Esbensen, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GlostrupUHNrct
Record Dates: First submitted 2024-07-04; First posted 2024-08-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Arthritis
Keywords: self-management; rheumatoid arthritis; axial spondyloarthritis; psoriatic arthritis; newly diagnosed; heiQ; quality of life
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Axial Spondyloarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: Randomization, allocation, and blinding Randomization 1:1 will be performed after baseline assessments and conducted using a computerized random number generator algorithm by the project manager. Randomization will be stratified by site. Therefore, a customized randomization table will be uploaded for each site to REDCap (Research Electronic Data Capture).
  The project manager will enroll participants and inform them whether they have been allocated to the intervention group or the control group (see Fig. 2 for participants flow through the trial). For participants randomized to the intervention group, the first individual session will be scheduled as soon as possible after allocation.
  Due to the character of the intervention, it is not possible neither to blind participants to their allocated intervention nor to blind the HP delivering the intervention. Analysis of data will be performed blinded to group allocation.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the NISMA intervention blinding of participants is impossible. However, the outcome assessor will be blinded, and participants will be asked not to disclose their group to the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlgroup (No Intervention): There are no established standards for identifying and addressing self-management needs in rheumatology outpatient consultations. Participants allocated to the control group will receive usual care, which consists of planned sessions with a rheumatologist and occasionally a nurse, a physiotherapist, and an occupational therapist. Those who started DMARDs of any type had an appointment with a nurse and a follow-up phone call. All participants will have the possibility to contact the outpatient clinic and talk to a nurse. Participants in the control group will be encouraged to maintain their usual daily routines and self-management practices until the follow-up assessment is conducted.
- intervention group (Experimental): Participants allocated to the intervention group will receive the NISMA Intervention in addition to usual care.
  Interventions: Behavioral: Newly diagnosed with Inflammatory arthritis - a Self-MAnagement intervention (NISMA)

INTERVENTIONS:
Behavioral: Newly diagnosed with Inflammatory arthritis - a Self-MAnagement intervention (NISMA) — The NISMA intervention is a flexible intervention and comprises three mandatory individual sessions with a nurse, supplemented by two optional group sessions over a period of 12 months, to provide comprehensive support tailored to each participant's needs. The intervention is grounded in the theoretical framework Social Cognitive Theory and inspired by the questioning techniques in Acceptance and Commitment Therapy (ACT). These methods play a crucial role in helping participants enhance their self-efficacy. The key components of our approach include: a person-centered approach by addressing challenges identified by each participant to foster self-efficacy through targeted problem-solving and goal-setting. This is utilized by interviewing techniques derived from ACT to assist participants in accepting and committing to self-management. The program is designed to last between 6-12 months, allowing for gradual skill development and adaptation.
  Arms: intervention group

SUMMARY:
Background:

In patients newly diagnosed with inflammatory arthritis, a self-management intervention is anticipated to enhance self-management skills, thereby improving patient function, well-being, and survival. The primary objective of the trial is to investigate the short-term efficacy of the NISMA intervention and usual care, compared to usual care alone (control group), on self-management skills and techniques in patients newly diagnosed with inflammatory arthritis.

Method:

This study aims to test the efficacy of the "Newly diagnosed with Inflammatory arthritis - a Self-MAnagement intervention" (NISMA) through a multicenter pragmatic randomized controlled trial (RCT). The trial will involve 130 patients newly diagnosed with IA from three Danish hospitals. Participants will be randomly assigned to either the NISMA intervention group or a control group receiving usual care. The NISMA intervention includes three mandatory individual sessions with a nurse, supplemented by two optional group sessions over 12 months.

Primary outcomes will be measured using the Health Education Impact Questionnaire (heiQ), focusing on the "skill and technique acquisition" domain. Secondary outcomes include other heiQ domains, quality of life, loneliness, physical function, pain intensity, pain, self-efficacy, anxiety and depression, fatigue, patient global assessment, disease activity, and medication adherence. Data will be collected at baseline, 12 months, and 18 months post-baseline.

Discussion:

This RCT will provide essential insights into the effectiveness of a targeted self-management intervention for patients newly diagnosed with IA. The NISMA intervention, developed following the Medical Research Council Framework for complex interventions, aims to improve self-management skills and overall QoL. By addressing the unique challenges faced by newly diagnosed patients, this study seeks to enhance the initial management of IA, aligning with the European Alliance of Associations for Rheumatology (EULAR) recommendations for self-management support. If successful, the NISMA intervention could represent a significant advancement in the non-pharmacological management of IA, offering a comprehensive, patient-centered approach that addresses both physical and psychological needs.

DETAILED DESCRIPTION:
Background:

Inflammatory arthritis (IA), including rheumatoid arthritis (RA), psoriatic arthritis (PsA), and axial spondyloarthritis (axSpA), encompasses acute and chronic joint diseases characterized by joint pain, swelling, and tenderness due to inflammation. IA affects over 2% of the global population, with significant variability. It can occur at any age and affects both sexes, with an etiology involving genetic and lifestyle factors. IA primarily causes joint pain and stiffness but can also impact other connective tissues. Without adequate treatment, IA can lead to functional decline, irreversible joint damage, comorbidities, and increased mortality. Early treatment with disease-modifying anti-rheumatic drugs (DMARDs) improves outcomes, with about 60% of RA patients achieving long-term remission. However, symptoms may persist and fluctuate, causing ongoing physiological and psychological distress, impacting daily activities and quality of life (QoL), even in remission.

Newly diagnosed patients with IA face particular challenges, including regular blood tests, lifelong medication, side effects, pain, fatigue, sleep disturbances, and increased risk of comorbidities like depression and cardiovascular disease. They often experience changes in body image, family, work, and social life. A crucial but often lacking aspect of IA care is empowering patients with a thorough understanding of their condition and effective self-management skills. Studies show that newly diagnosed patients benefit from regular consultations and support from health professionals (HPs) to manage the physical, emotional, and social impacts of IA. Enhanced self-management, defined as the ability to manage symptoms, treatments, and lifestyle changes, can improve QoL in chronic illness patients. EULAR recommends incorporating self-management into daily rheumatology care, including patient education and key approaches like problem-solving and action planning. Despite this, no IA-specific self-management interventions focused on newly diagnosed patients exist.

Rationale:

To address this gap, the "Newly diagnosed with Inflammatory arthritis - a Self-MAnagement intervention" (NISMA) was developed. Following the Medical Research Council (MRC) Framework [29,30] for developing and evaluating complex interventions, the researchers developed NISMA and tested its feasibility and fidelity. Feedback from patients and HPs led to adjustments in session duration, the number of sessions, flexible scheduling, recruitment strategies, and inclusion criteria for axSpA patients. Group sessions were made optional, and more emphasis was placed on certain behavior change techniques.

The hypothesis is that the adapted NISMA intervention will surpass usual care in enhancing self-management skills. The next step is to test this hypothesis in a randomized controlled trial (RCT). If effective, a cost-effectiveness analysis will be conducted.

Objectives:

The primary objective of this trial is to investigate the short-term efficacy of the NISMA intervention and usual care, compared to usual care alone, on "self-management skills and techniques" in patients newly diagnosed with inflammatory arthritis, from baseline to completion of the intervention (after 12 months).

Our key secondary objectives are to compare the short-term efficacy of the NISMA intervention, relative to usual care on self-management skills, quality of life, loneliness, physical function, pain intensity, pain self-efficacy, anxiety and depression, fatigue, patient global assessment, disease activity, C-reactive protein (CRP), and medication adherence from baseline to completion of the intervention (after 12-months).

Other objectives are to test the longer-term efficacy of the intervention relative to usual care, on self-management skills, quality of life, loneliness, physical function, pain intensity, pain self-efficacy, anxiety and depression, fatigue, patient global assessment, disease activity, C-reactive protein (CRP), and medication adherence at follow-up 18-months after baseline.

Trial design:

The trial is designed as a multicenter pragmatic randomized trial with a two-group parallel design in a superiority framework. Participants will be allocated in a 1:1 ratio; after providing informed consent and completing baseline assessments, they will be randomized to either the NISMA intervention (experimental group) or usual care (control group) with no protocolized treatment.

Setting:

Patients will be included from the following centers: the Center for Rheumatology and Spine Diseases, Rigshospitalet University Hospital, Copenhagen, and department of Rheumatology and Spine Diseases, Holbæk Hospital; both in Denmark.

Sample size and power calculation:

As no established thresholds exist for clinically relevant changes in heiQ domains, we refer to prior research [61,62]. In the skills acquisition domain, we found mean differences between groups ranging from 0.22 to 0.38. Therefore, we decided that a minimal important difference probably corresponds to a target difference of 0.30 with a standard deviation (SD) of 0.55 for the heiQ 'skill and technique acquisition' domain (primary endpoint) from baseline to 12 months after baseline. To achieve a statistical power of 80% and a significance level set at an alpha of 0.05, our calculations indicated a need for 54 patients per group (i.e., enrolling 108 patients in the ITT Population). Incorporating an anticipated dropout rate of 15% from our feasibility study, the sample size would correspond to 127. Consequently, we revised the necessary sample size to approximately 65 patients per group (i.e., 130 patients in the ITT population) to achieve a reasonable statistical power to identify a statistically significant difference between the intervention and control group (i.e., corresponding to a statistical power of 87% in the best-case scenario).

Statistical Methods:

Descriptive statistics for baseline data will be reported in a Table 1 format; reported separately for each treatment group. These descriptive statistics will summarize the characteristics of participants at baseline, including demographic information and outcome variables relevant to the trial. Descriptive statistics include the mean and standard deviation (SD), or median and interquartile ranges (if applicable). For categorical data we will report the count and percentages.

The main analyses will be based on the Intention to Treat (ITT) population, i.e., including all randomized patients with a baseline measure available [63]. The ITT principle asserts the effect of a treatment policy (that is, the planned treatment regimen), rather than the actual treatment given (i.e., it is independent of treatment adherence) [9]. Accordingly, participants allocated to a treatment group (NISMA and Control, respectively) will be followed up, assessed, and analyzed as members of that group, irrespective of their adherence to the planned course of treatment (i.e., independent of withdrawals and cross-over phenomena).

All 95% confidence intervals and P values will be two-sided. We will not apply explicit adjustments for multiplicity, rather we will analyze the key secondary outcomes and interpret these as endpoints in a prioritized order (e.g., "gatekeeping procedure"): The analyses of the secondary endpoints will be performed and interpreted in sequence until one of the analyses fails to show the statistically significant difference, or until all analyses have been completed at a statistical significance level of 0.05 (P<0.05). All analyses in the statistical hierarchy will be based on the treatment policy estimand (the primary estimand, i.e., the ITT principle), which quantifies the average treatment effect regardless of adherence to treatment or initiation of rescue interventions between baseline and month 12.

The primary endpoint will be based on the change in heiQ from baseline to 12 after baseline, estimated as the difference between least squares means. In our main analyses, estimations of between-group differences for all continuous outcomes will be conducted after 12 months.

Continuous outcome measures will be analyzed using analysis of covariance, with randomized treatment, trial site, and type of IA diagnoses as factors, and baseline (pre-exposure) value as a covariate. Categorical endpoints will be analyzed using logistic regression, with the same factors and covariates. A multiple imputation approach will be used in which missing data are imputed from month 12 measurements from participants in the same treatment group. A series of complete data sets will be generated and analyzed, and the results will be combined using the Rubin formula [64] to obtain overall estimates. While binary outcomes will be analyzed and initially reported using Odds Ratios with 95%confidence intervals (95%CIs), all between-group differences 95%CIs for continuous outcomes will be based on the least-square means, adjusted for baseline levels and stratifying factors to minimize random variation [65].

Project Group:

The project group includes two patient research partners, professors in rheumatology, nursing, epidemiology, and postdocs in occupational therapy and nursing. They bring expertise in RCTs, qualitative research, and epidemiology.

Patient Involvement:

Three patients were involved in the initial design and development of the NISMA intervention. During feasibility testing, patients were interviewed to include their views. A patient with RA serves as a research partner, ensuring the patient perspective is maintained throughout the project [54].

Dissemination and Protocol Amendments:

Results will be disseminated through peer-reviewed journals, academic conferences, news outlets, social media, multimedia materials, and popular science magazines. Authorship will follow ICMJE guidelines. Any significant protocol modifications will be communicated to the Committee on Health Research Ethics for The Capital Region of Denmark, registered on ClinicalTrials.gov, and detailed in the primary RCT report.

Discussion:

This trial addresses the need for targeted interventions for newly diagnosed IA patients. By enhancing self-management skills early, better long-term outcomes are anticipated. The NISMA RCT aims to evaluate the effectiveness of a targeted self-management intervention. Developed through a feasibility study and process evaluation, the intervention is tailored to newly diagnosed patients and may prove more effective than previous interventions.

The trial aligns with EULAR's emphasis on high-quality, systematic, and personalized care in rheumatology. Educating health professionals in group facilitation, problem-solving, goal-setting, and cognitive-behavioral techniques could enhance multidisciplinary collaboration and patient satisfaction. If effective, a cost-effectiveness analysis will follow, focusing on integrating the intervention into clinical practice.

Limitations:

The main limitations are the inability to blind participants, potential spillover effects, variability in usual care, and the individually adjusted intervention content. However, outcome assessors will be blinded, and participants will be instructed not to disclose their group.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they are adults aged 18 years or older with one of the following conditions:

* Rheumatoid Arthritis (RA) with ICD-10 codes: M05.3, M05.9, M05.8, M06.9 diagnosed within the last 6 months
* Psoriatic Arthritis (PsA) with ICD-10 codes: M073.A, M073.B diagnosed within the last 6 months
* Axial Spondyloarthritis (axSpA) with ICD-10 codes: M45.9, M46.1, M46.8, M46.9, diagnosed within the last 12 months, and has initiated biological treatment

Patients with axSpA will have unique inclusion criteria due to NSAIDs being the first-line pharmacological treatment. For those effectively treated with NSAIDs and exercise, treatment is transitioned to their general practitioner. Therefore, only those who have initiated biological treatment will be included.

Exclusion Criteria:

Patients will be excluded if they:

* have insufficient language skills to discuss the topics in the intervention in Danish
* are receiving chemo-therapy treatment for malignancies
* are pregnant
* have severe mental illness.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome and endpoint | Baseline-end of intervention (12 months after baseline).
  The primary outcome measure is self-management skills, assessed by the Health Education Impact Questionnaire (heiQ) - the skill and technique acquisition domain. (Higher score is better). The primary endpoint will be the difference in least squares means between groups, analyzed at 12 months from baseline.

SECONDARY OUTCOMES:
Self-management skills measured by the Health Education Impact Questionnaire (heiQ) | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  heiQ domains: health-directed activity; positive and active engagement in life; emotional wellbeing; self-monitoring and insight; constructive attitudes and approaches; social integration and support. (Higher score is better). The corresponding endpoints is the between-group difference in least squares means from the 6 heiQ domains after 12 months. Endpoints in the extension study are the between-group difference in least squares means in heiQ domain 1, 2, 3, 4, 5, 6, 7, and 8 after 24 months.
Health Related Quality of Life | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  Health Related Quality of Life measured by European Quality of Life (EQ5D). (Higher score is better). The corresponding endpoint is the between-group difference in least squares means from EQ5D-5L after 12 months. Endpoint in the extension study is between group difference in EQ5D-5L 24 months after baseline.
Loneliness | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  Loneliness will be measured by The Three Item Loneliness Scale ( 3 categories, higher score is worse). The corresponding endpoint is the between-group difference after 12 months. Endpoint in the extension study is between group difference 24 months after baseline.
Physical function | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  Physical function measured by Modified Health Assessment Questionnaire (MHAQ). (Higher score is worse). The corresponding endpoint is the between-group difference in least squares means from MDHAQ after 12 months. Endpoint in the extension study is between group difference in MDHAQ 24 months after baseline.
Pain Intensity | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  Pain Intensity measured by VAS (0-100). (Higher score is worse). The corresponding endpoint is the between-group difference in least squares means from VAS after 12 months. Endpoint in the extension study is between group difference in VAS 24 months after baseline.
Pain self-efficacy | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  Pain self-efficacy measured by the Arthritis specific Self-Efficacy measurement tool (ASES-pain). (Higher score is better). The corresponding endpoint is the between-group difference in least squares means from ASES-pain after 12 months. Endpoint in the extension study is between group difference in ASES-pain 24 months after baseline.
Fatigue | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  Fatigue measured by the Bristol Rheumatoid Arthritis Fatigue Numeric Rating Scale (BRAF-NRS). (Higher score is worse). The corresponding endpoint is the between-group difference in least squares means from BRAF-NRS after 12 months. Endpoint in the extension study is between group difference in BRAF-NRS 24 months after baseline.
Fatigue | Baseline-end of intervention (12 months after baseline), and 24 months after baseline.
  VAS-fatigue (0-100). (Higher score is worse). The corresponding endpoint is the between-group difference in least squares means from VAS after 12 months. Endpoint in the extension study is between group difference in VAS 24 months after baseline.
Patient global | Baseline-end of intervention (12 months after baseline), and 24 months after baseline
  Patient global assessment measured by VAS-Global. (Higher score is worse). The corresponding endpoint is the between-group difference in least squares means from VAS after 12 months. Endpoint in the extension study is between group difference in VAS 24 months after baseline.
Disease activity | Baseline-end of intervention (12 months after baseline), and 24 months after baseline
  Disease activity will be measured by composite scores depending on the rheumatic diagnoses. For RA: Disease Activity Score in 28 joints (DAS28), for axSpA: the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), and for PsA: the Disease Activity index for Psoriatic Arthritis (DAPSA). (Higher score is worse).
Medication adherence | Baseline-end of intervention (12 months after baseline), and 24 months after baseline
  Medication adherence will be measured by the Compliance Questionnaire Rheumatology (CQR)-5-item scale. (Higher score is better). The corresponding endpoint is the between-group difference in least squares means from CQR after 12 months. Endpoint in the extension study is between group difference in CQR 24 months after baseline.
Anxiety and depression | Baseline-end of intervention (12 months after baseline), and 24 months after baseline
  Anxiety and depression will be measured by the Hospital Anxiety and Depression Scale (HADS). (higher score is worse). The corresponding endpoint is the between-group difference in least squares means from HADS after 12 months. Endpoint in the extension study is between group difference in HADS 24 months after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Bente A Esbensen, Principal Investigator — Rigshospitalet, Glostrup, Center for Rheumatology and Spine Diseases. COPECARE
Locations (2):
- Denmark (2):
  - Rigshospitalet, Center for Rheummatology and Spine Diseases, Glostrup Municipality
  - Holbæk sygehus, Holbæk

IPD SHARING:
Plan to Share IPD: No
The dataset includes potentially identifiable or sensitive data, which, if disclosed publicly, could jeopardize the participants' privacy. Consequently, in compliance with the regulations established by the Danish Data Protection Agency, the data is not accessible to the public. However, interested parties may obtain access by making a reasonable request to the corresponding author.

REFERENCES:
- [Derived] Lindgren LH, Thomsen T, Hetland ML, Aadahl M, de Thurah A, Christensen R, Esbensen BA. Effect of a self-management intervention for newly diagnosed inflammatory arthritis: study protocol for a randomized controlled trial. Trials. 2025 Nov 27;26(1):594. doi: 10.1186/s13063-025-09192-z. PMID 41310759

DOCUMENTS (2):
  • Study Protocol (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT06533423/Prot_000.pdf
  • Statistical Analysis Plan (2026-02-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT06533423/SAP_001.pdf